CLINICAL TRIAL: NCT03224910
Title: Diagnostic Efficiency of Needle Core Biopsy Touch Imprints Versus Fine Needle Aspiration Smears at the Time of Rapid on Site Interpretation
Brief Title: Diagnostic Efficiency of Touch Imprints Versus Smears
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Maria F. Gonzalez, Assistant Professor of the department of pathology, University of Mississippi Medical Center
Other Study IDs: 2017-0076
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Diagnostic Self Evaluation
Keywords: FNA, smears, imprints, ROSE

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cytologic techniques used for rapid on site interpretation — Diagnostic efficiency of touch imprints of needle core biopsies vs smears of fine needle aspirations during rapid on-site interpretation

SUMMARY:
Cytopathologists work along with radiologist in the diagnosis of lesions. Rapid on site interpretation (ROSE) of fine needle aspiration (FNA) smears of radiologically suspicious lesions is a common clinical practice. In the last years, the investigators have seen trend towards needle core biopsies of radiologically suspicious lesions. The investigators want to analyze the challenges of rapid on site interpretation of touch imprints (TI) of needle core biopsies (NCB) versus fine needle aspiration smears.

DETAILED DESCRIPTION:
This is a retrospective study in which the investigators will analyze the quality of the smears and the touch imprints, the cellularity, the cytomorphologic features of the specimens and the presence of adequate material for ancillary studies. The specimens will be searched through the University of Mississippi Medical Center's Pathology Laboratory information system (Copath), from January 2011 to December 2017. The retrospective cases (January 2011 up to now) will be retrieved using natural language search of fine needle aspiration and touch imprints. The slides of those cases will be reviewed and the cytomorphologic features will be described.

ELIGIBILITY:
Inclusion Criteria:

* 1. Computerized tomography (CT)-Guided Fine needle aspiration (FNA) /Needle core biopsy (NCB) specimens from any site.2. Ultrasound (US) guided FNA/NCB.

Exclusion Criteria:

* 1. Specimens obtained through endoscopic fine needle aspirations.2. US-guided specimens from thyroid3. Exfoliative specimens like sputum or urine4. Gynecologic cytology specimens.5. Outside cytology consult cases6. Pathologist performed FNA's

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patient that has required a fine needle aspiration or needle core biopsy at UMMC to diagnose a lesion regardless of the age, sex or any other condition.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Number of cases with enough diagnostic features on the FNA smears and/or touch imprints of NCB. | January 2011 to December 2017
  All the cytology cases with rapid on site examination (ROSE) of FNA smears and/or touch imprints of needle core biopsies from January 1st/2011 to December 31st/ 2017, will be retrieved using the University of Mississippi Medical Center's Pathology Laboratory information system (Copath). The investigators will review the cases and get a number of cases with enough diagnostic features (based on the cytomorphologic features of the cells, quality of the smears and touch imprints, and the cellularity) on each case.

CONTACTS AND LOCATIONS:
Overall Officials: Maria F Gonzalez, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta NJ, Wang HH. Increase of core biopsies in visceral organs--experience at one institution. Diagn Cytopathol. 2011 Nov;39(11):791-5. doi: 10.1002/dc.21456. Epub 2010 Oct 19. PMID 20960472
- [Result] Aisner DL, Sams SB. The role of cytology specimens in molecular testing of solid tumors: techniques, limitations, and opportunities. Diagn Cytopathol. 2012 Jun;40(6):511-24. doi: 10.1002/dc.22820. PMID 22619126
- [Result] Padmanabhan V, Barkan G, and Nayar R. Cytopathology + More | Assessing needle core biopsy adequacy-survey of practices. http://www.captodayonline.com/assessing-needle-core-biopsy-adequacy-survey-practices-516/
- [Result] Rekhtman N, Kazi S, Yao J, Dogan S, Yannes A, Lin O, Silk M, Silk T, Durack JC. Depletion of Core Needle Biopsy Cellularity and DNA Content as a Result of Vigorous Touch Preparations. Arch Pathol Lab Med. 2015 Jul;139(7):907-12. doi: 10.5858/arpa.2014-0392-OA. Epub 2014 Dec 18. PMID 25521802
- [Result] Dogan S, Becker JC, Rekhtman N, Tang LH, Nafa K, Ladanyi M, Klimstra DS. Use of touch imprint cytology as a simple method to enrich tumor cells for molecular analysis. Cancer Cytopathol. 2013 Jul;121(7):354-60. doi: 10.1002/cncy.21292. Epub 2013 Apr 10. PMID 23576371
- [Result] Mangia A, Chiriatti A, Chiarappa P, Incalza MA, Antonaci G, Pilato B, Simone G, Tommasi S, Paradiso A. Touch imprint cytology in tumor tissue banks for the confirmation of neoplastic cellularity and for DNA extraction. Arch Pathol Lab Med. 2008 Jun;132(6):974-8. doi: 10.5858/2008-132-974-TICITT. PMID 18517281
- [Result] Hahn PF, Eisenberg PJ, Pitman MB, Gazelle GS, Mueller PR. Cytopathologic touch preparations (imprints) from core needle biopsies: accuracy compared with that of fine-needle aspirates. AJR Am J Roentgenol. 1995 Nov;165(5):1277-9. doi: 10.2214/ajr.165.5.7572518.
- [Result] Chandan VS, Zimmerman K, Baker P, Scalzetti E, Khurana KK. Usefulness of core roll preparations in immediate assessment of neoplastic lung lesions: comparison to conventional CT scan-guided lung fine-needle aspiration cytology. Chest. 2004 Sep;126(3):739-43. doi: 10.1378/chest.126.3.739. PMID 15364750